CLINICAL TRIAL: NCT03707236
Title: The Use of Teledermatology in the Treatment of Patients With Severe Acne on Isotretinoin: A Randomized-controlled Trial
Brief Title: The Use of Teledermatology in the Treatment of Patients With Severe Acne on Isotretinoin
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Study was planned prior to COVID-19; after pandemic teledermatology use became prevalent making the results of this study no longer necessary/relevant
Sponsor: Massachusetts General Hospital (Other)
Responsible Party: Principal Investigator, Daniela Kroshinsky, Director of Inpatient Dermatology, Associate Professor of Dermatology, Massachusetts General Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: 2018P001749
Record Dates: First submitted 2018-09-28; First posted 2018-10-16 (Actual); Last update posted 2023-04-06 (Actual); Status verified 2023-04

CONDITIONS: Acne Vulgaris
Keywords: Isotretinoin
MeSH Terms: conditions — Acne Vulgaris

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Treatment arm (Experimental): Patients in the treatment arm will have monthly office visits for weeks 0-4 and then have monthly teledermatology visits during weeks 8-20 with a final office visit at week 24. Standardized baseline photographs including 3 facial images (front, left, and right) as well as 2 truncal images of the chest and back (if affected) will be taken in the office at treatment week 0 and 24 for all patients. All patients will be required to take photos in front of a white wall to facilitate blinding.
  Interventions: Behavioral: Teledermatology visits
- Control arm (No Intervention): Patients in the control arm will have the same series of photographs taken at each monthly visit. These patients will also be required to fill out a monthly survey assessing acne severity, quality of life, cost of attending appointment, time missed from school/work, satisfaction with treatment (only to be reviewed by study staff) and will be screened for adverse events by their provider. Every patient will be counseled about isotretinoin and contraception (if applicable) by their provider in order to adhere with iPledge requirements. All photographs will be uploaded into the patient's medical record. The physician will be required to document a progress note in the electronic medical record after each visit as per standard hospital protocol.

INTERVENTIONS:
Behavioral: Teledermatology visits — Patients in the treatment arm will be taught by study staff how to take the standardized photos of themselves at treatment week 4 (prior to initiation of teledermatology visits). For patients in the treatment arm, the teledermatology visits will be managed by the study staff. A monthly teledermatology visit will consist of sending facial and truncal (if affected) clinical images to a the study staff using Patient Gateway. Once this is completed, the patient and a member of the study staff will have a scheduled telephone appointment during which the provider will screen for any adverse events and will provide counseling as outlined in iPledge guidelines. The patient will also be asked to verbally complete a monthly survey assessing acne severity, quality of life, cost attributable to the appointment, time missed from school/work, satisfaction with treatment. All photographs will be uploaded in LMR/EPIC in the patient's medical record.
  Arms: Treatment arm

SUMMARY:
This is a non-blinded randomized controlled non-inferiority trial designed to assess the efficacy and role of teledermatology visits in the treatment of patients with severe acne starting isotretinoin. Males and females 16 years or older will be randomized to either the control arm (monthly office visits during treatment weeks 8-20) or treatment arm (teledermatology visits during treatment weeks 8-20). The primary outcome is the change in total inflammatory lesion count. Secondary outcomes include changes in acne severity based on the Leeds scale, patient satisfaction, acne severity as perceived by the patient, cost and time-lost to patients and families, need for interim and unexpected urgent appointments, adverse medication effects. The investigators are hypothesizing that patients randomized to the treatment arm will have no statistically significant difference in total inflammatory lesion count or acne severity than the control arm. The investigators also hypothesize that adverse events will be equivalent in both groups and the treatment arm will report less cost associated with visits.

DETAILED DESCRIPTION:
The role of telemedicine in dermatology is ever-expanding. Currently, teledermatology has been shown to be advantageous in disease processes that require frequent office follow-up visits such as psoriasis. In 2010, Watkins et al. demonstrated that teledermatology was effective in treating patients 16 years and older with moderate acne and demonstrated equivocal clinical outcomes as traditional office visits along with equivocal patient and provider satisfaction scores. More recently, Fruhauf et al. conducted a small study examining patients with severe acne on isotretinoin and found similar results in terms of safety and efficacy. Patients with severe acne on isotretinoin therapy currently are scheduled for monthly office visits in the dermatology clinic for at least six consecutive months during which time the severity of their acne is assessed by a dermatologist and dose adjustments are made accordingly. Patients are also required to get monthly laboratory studies immediately before, during, or after their visit, and this must be reviewed by the provider prior to prescription renewal according to iPledge guidelines. Given the fact that this medication is typically prescribed to teenagers or young adults, the high frequency of office visits put a significant burden on both patients and their families and results in unnecessary time missed from work or school.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have a diagnosis of severe acne by a dermatologist with a plan of initiating treatment with isotretinoin
* Patients must first be enrolled in iPledge prior to eligibility

Exclusion Criteria:

* Patients who have baseline hepatic dysfunction or hypertriglyceridemia
* Patients with a history of depression, suicide attempts or suicidal ideation
* Patients without access to internet or a camera (including portable camera and/or smart phone) at home
* Patients who are pregnant - absolute contraindication

Min Age: 16 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2023-04-01 (Actual); Primary Completion 2023-04-01 (Actual); Study Completion 2023-04-01 (Actual)

PRIMARY OUTCOMES:
Change in total inflammatory lesion count | Up to 24 weeks
  Lesion counting involves counting the number of inflammatory lesions on the face, chest, or back. This excludes comedonal acne.

SECONDARY OUTCOMES:
Changes in acne severity | Up to 24 weeks
  The Leeds scale will be used to assess patients' acne, which examines the extent of inflammation, range and size of inflamed lesions, and associated erythema. The Leeds technique is a counting system for detailed work in therapeutic trials. A scale of 0 (no acne) to 10 (most severe) is used for grading.
Patient satisfaction | Up to 24 weeks
  This will be assessed by having the patient fill out a survey about how much time they missed and costs they may have incurred to go to the appointment. They will also be asked questions about how they feel their acne has affected their lives.

REFERENCES:
- [Background] Koller S, Hofmann-Wellenhof R, Hayn D, Weger W, Kastner P, Schreier G, Salmhofer W. Teledermatological monitoring of psoriasis patients on biologic therapy. Acta Derm Venereol. 2011 Oct;91(6):680-5. doi: 10.2340/00015555-1148. PMID 21879250
- [Background] Watson AJ, Bergman H, Williams CM, Kvedar JC. A randomized trial to evaluate the efficacy of online follow-up visits in the management of acne. Arch Dermatol. 2010 Apr;146(4):406-11. doi: 10.1001/archdermatol.2010.29. PMID 20404229
- [Background] Fruhauf J, Krock S, Quehenberger F, Kopera D, Fink-Puches R, Komericki P, Pucher S, Arzberger E, Hofmann-Wellenhof R. Mobile teledermatology helping patients control high-need acne: a randomized controlled trial. J Eur Acad Dermatol Venereol. 2015 May;29(5):919-24. doi: 10.1111/jdv.12723. Epub 2014 Sep 26. PMID 25258175
- [Background] Risk evaluation and mitigation strategy (REMS). iPLEDGE Program: Single Shared System for Isotretinoin. http://www.fda.gov/downloads/Drugs/DrugSafety/PostmarketDrugSafetyInformationforP atientsandProviders/UCM234639.pdf . Accessed November 11, 2012.
- [Background] Lucky AW, Barber BL, Girman CJ, Williams J, Ratterman J, Waldstreicher J. A multirater validation study to assess the reliability of acne lesion counting. J Am Acad Dermatol. 1996 Oct;35(4):559-65. doi: 10.1016/s0190-9622(96)90680-5. PMID 8859284
- [Background] Bergman H, Tsai KY, Seo SJ, Kvedar JC, Watson AJ. Remote assessment of acne: the use of acne grading tools to evaluate digital skin images. Telemed J E Health. 2009 Jun;15(5):426-30. doi: 10.1089/tmj.2008.0128. PMID 19548822
- [Background] Burke BM, Cunliffe WJ. The assessment of acne vulgaris--the Leeds technique. Br J Dermatol. 1984 Jul;111(1):83-92. doi: 10.1111/j.1365-2133.1984.tb04020.x. PMID 6234917
- [Background] Lee YH, Scharnitz TP, Muscat J, Chen A, Gupta-Elera G, Kirby JS. Laboratory Monitoring During Isotretinoin Therapy for Acne: A Systematic Review and Meta-analysis. JAMA Dermatol. 2016 Jan;152(1):35-44. doi: 10.1001/jamadermatol.2015.3091. PMID 26630323
- [Background] Suneja T, Smith ED, Chen GJ, Zipperstein KJ, Fleischer AB Jr, Feldman SR. Waiting times to see a dermatologist are perceived as too long by dermatologists: implications for the dermatology workforce. Arch Dermatol. 2001 Oct;137(10):1303-7. doi: 10.1001/archderm.137.10.1303. PMID 11594853
- [Background] Tsang MW, Resneck JS Jr. Even patients with changing moles face long dermatology appointment wait-times: a study of simulated patient calls to dermatologists. J Am Acad Dermatol. 2006 Jul;55(1):54-8. doi: 10.1016/j.jaad.2006.04.001. Epub 2006 May 6. PMID 16781292